CLINICAL TRIAL: NCT05231447
Title: Registry of Congenital Anomalies in Nouvelle-Aquitaine, France
Brief Title: Birth Defect Registry in South West Region of France
Acronym: ATENA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut de Recherche en Santé Publique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/36
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Congenital Abnormalities
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Environmental survey — Exposure to environmental factors, drugs or individual toxicity during the periconceptional period and at the beginning of the pregnancy will be investigated by means of a questionnaire administered to the parents. This questionnaire, drawn up by the "Aquitaine Reproduction Enfance Maternité et Impact Santé-environnement" (ARTEMIS) centre and completed by both members of the couple, will constitute an initial assessment that will make it possible to collect environmental exposures for the parents of cases identified by the register.

SUMMARY:
Regional population-based registry for the epidemiological surveillance of congenital anomalies

DETAILED DESCRIPTION:
By systematically collecting data on congenital anomalies, the registry aims to :

* provide essential epidemiological information on congenital anomalies in South West of France
* Promote etiological research concerning congenital anomalies, particularly with regard to environmental risk factors (systematic questionnaire) and other teratogenic agents (drugs)
* act as an information and resource center for the population, health professionals and managers regarding clusters or exposures or risk factors of concern.
* evaluate the effectiveness of primary prevention
* assess the impact of developments in prenatal screening
* study the fate of children with congenital anomalies, particularly in terms of neurodevelopment, through the creation of cohorts.

ELIGIBILITY:
Inclusion Criteria:

Children or Fetuses:

* Born alive or stillborn or fetal death in utero or medical termination of pregnancy
* Of mothers domiciled in New Aquitaine at the time of delivery
* And presenting a congenital or chromosomal anomaly defined according to the EUROCAT network, diagnosed antenatally or postnatally up to one year of life.
* Of which the non-opposition of both holders or of the only holder of parental authority has been given
* Whose mother and/or father is affiliated or beneficiary of a social security system.

Exclusion Criteria:

* Refusal of at least one of the holders of parental authority

Ages: 1 Minute to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cases are defined as all fetuses/children under 1 year of age with a congenital or chromosomal abnormality as defined by the european surveillance of congenital anomalies (EUROCAT) network.
  The excluded minor anomalies are established by EUROCAT. The register covers the geographical area of the Nouvelle Aquitaine region in France.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of congenital anomalies | 1 year-old

SECONDARY OUTCOMES:
Measure of the incidence of congenital anomalies in south west region of France | 1 year-old
  In number of new cases, expected 2500 cases/year
Identification of environmental factors associated with congenital anomalies | 1 year-old
  Environment related variables and drug exposure before (father and mother) and during pregnancy (mother)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Thomas-Chabaneix, MD, Principal Investigator — University Hospital, Bordeaux; Marianne Saves, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France